CLINICAL TRIAL: NCT01521715
Title: A Single Arm Multicentre Study Evaluating Pazopanib in First-line Treatment of Poor-risk Patients With Locally Advanced or Metastatic Renal Cell Carcinoma
Brief Title: First Line Pazopanib in Poor Risk Patients With Metastatic Renal Cell Carcinoma
Acronym: FLIPPER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: iOMEDICO AG (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iOM-605; 2011-001138-40 (EudraCT Number)
Record Dates: First submitted 2011-12-21; First posted 2012-01-31 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Locally Advanced and/or Metastatic Renal Cell Carcinoma; Carcinoma, Renal Cell; Clear-cell Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Clear-cell metastatic renal cell carcinoma | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pazopanib (Experimental): 800 mg (2x400mg) pazopanib per day
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — 800 mg (2x400mg) pazopanib per day should be taken orally without food at least one hour before or two hours after a meal until progression or occurrence of intolerable toxicity.
  Other Names: Votrient

SUMMARY:
Patients with advanced renal cell carcinoma (RCC) are classified according to Memorial Sloan-Kettering Cancer Center (MSKCC) criteria in three risk-groups: favourable, intermediate and poor. To our knowledge there is only one study which examined the poor risk group (Hudes et al.), which led to the approval of temsirolimus in this population. However temsirolimus demonstrated a low response rate of 8.6% according to Response Evaluation Criteria In Solid Tumor (RECIST) criteria and a Progression free Survival (PFS) of 5.5 months and not all patients are suitable for temsirolimus treatment.

Thus, in clinical routine high-risk patients are also treated with multi Tyrosinkinase Inhibitors (mTKI). To date, a prospective data acquisition and control of effectiveness of a mTKI-treatment in high-risk patients has not been conducted.

Pazopanib was recently approved for the first-line treatment of advanced renal cell carcinoma in Europe and the USA. In the pivotal Phase III trial only nine patients in the pazopanib group were poor risk according to MSKCC risk criteria and no analysis of this subgroup was performed. Therefore further data in this group of patients with high medical need is needed.

Currently there are no well-established predictive or prognostic biomarkers in RCC-mTKI treatment. This is one of the most important scientific questions in this field. In addition to the clinical endpoints in this study, the comprehensive biomarker program seeks to evaluate biomarker candidates and will help to learn more about the effects of pazopanib on the human organism.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic or locally advanced (defined as non operable tumor), predominantly clear cell renal cell carcinoma.
* At least three of the following five predictors of short survival are required:

  * Lactate Dehydrogenase (LDH) > 1.5 x Upper Limit of Normal (ULN)
  * Hemoglobin < Lower Limit of Normal (LLN)
  * corrected serum calcium level > 10 mg/dl (2.5 mmol/l)
  * time from initial diagnosis of renal-cell carcinoma to occurrence of metastases of less than 1 year
  * Karnofsky Status of 60 or 70
* Karnofsky Status ≥ 60
* Age ≥ 18 years or legal age of consent if greater than 18 years
* Dated and signed written informed consent prior to performance of study-specific procedures or assessments
* Patients with at least one measurable disease, as defined by RECIST 1.1
* Fresh or archived tumor tissue should be provided for all subjects for biomarker analysis before or during treatment with pazopanib.
* Adequate organ system function as defined as:
* Subjects may not have had a transfusion within 7 days of screening assessment.
* Subjects receiving anticoagulant therapy are eligible if their International Normalized Ratio (INR) is stable and within the recommended range for the desired level of anticoagulation.
* Concomitant elevations in bilirubin and aspartate aminotransferase (AST) or alanine aminotransferase (ALT) above 1.0 x ULN are not permitted. Patients with Gilbert's disease and elevation of indirect bilirubin only can be considered like patients with normal bilirubin.
* Compliance of the patient

Exclusion Criteria:

* Other malignancy. (Patients who have undergone prior radical or partial nephrectomy for RCC are allowed). Subjects who have had another malignancy and have been disease-free for five years, or subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible.
* Prior systemic treatment for renal cell carcinoma. (NB: all treatments, neo-adjuvant, adjuvant or for locally advanced or metastatic RCC are not permitted.)
* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for 6 months prior to first dose of study drug. Screening with CNS imaging studies (computed tomography (CT) or magnetic resonance imaging (MRI) is required only if clinically indicated or if the subject has a history of CNS metastases.
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to: Malabsorption syndrome, major resection of the stomach or small bowel.
* Presence of uncontrolled infection (> grade 2 NCI-CTCAE Version 4.03).
* Corrected QT interval (QTc) > 480 msecs using Bazett's formula
* History of any one or more of the following cardiovascular conditions within the past 6 months:

  * Myocardial infarction
  * Cardiac angioplasty or stenting
  * Unstable angina
  * Coronary artery bypass graft surgery
  * Symptomatic peripheral vascular disease
  * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
* Poorly controlled hypertension
* History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months. Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible
* Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer.
* Evidence of active bleeding or bleeding diathesis.
* Known endobronchial lesions or lesions infiltrating major pulmonary vessels
* Hemoptysis in excess of 2.5 ml (or one half teaspoon ) within 8 weeks prior to first dose of study drug
* Any serious or unstable pre-existing medical, mental, or other condition, medical, social or mental impairment or drug abuse that could comprise or interfere with the subject's safety, provision of informed consent, or compliance to study procedures.
* Unable or unwilling to discontinue use of prohibited medications for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study.
* Simultaneous participation in another clinical drug study
* Known infection with Human Immunodeficiency Virus (HIV) or chronic hepatitis B or C
* Pregnant or breast-feeding women. Female subjects of childbearing potential need to be negatively tested prior and as close to the start of therapy as possible, at least within 14 days. Women participating in this trial are required to use adequate contraception. Female subjects who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug
* Subjects who are unable to take oral medication
* Known hypersensitive reaction to any of the components of study treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-01-24 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Rate of poor risk patients as defined by the Memorial Sloan-Kettering Cancer Center (MSKCC) criteria who are free of disease progression at 6 months after start of first line treatment with pazopanib. | from registration until progression of disease or death, assessed up to 6 months

SECONDARY OUTCOMES:
Overall survival of poor risk patients treated with pazopanib. | from registration until death of any cause assessed up 24 months
Number, characteristics and severity of Adverse Events | from first dose of pazopanib until 30 days after last dose, death or end of study, whichever came first
Progression free survival of patients treated with pazopanib | From date of registration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 20 months
Overall response rate and duration of response according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 | From date of registration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 20 months
Relation between biomarkers and clinical outcome (response, stable disease, progression of disease) | From date of registration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 20 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Staehler, PD MD, Principal Investigator — Ludwig-Maximilians-Universität München, Klinikum Grosshadern
Locations (8):
- Germany (8):
  - Urolog. Klinik im Waldkrankenhaus St. Marien, Friedrich-Alexander-Universität, Erlangen
  - Universitätsklinikum Essen, Klinik f. Urologie, Essen
  - Med. Klinik II, Johann-Wolfgang-Goethe-Universität, Frankfurt
  - Medizinisches Versorgungszentrum (MVZ) Osthessen GmbH, Fulda
  - Universitätsmedizin Greifswald, Greifswald
  - Medizinische Hochschule Hannover, Hanover
  - Ludwig-Maximilians-Universität (LMU) München, Klinikum Grosshadern, München
  - Universitätsklinikum Münster, Münster

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Staehler M, Panic A, Goebell PJ, Merling M, Potthoff K, Herrmann E, de Geeter P, Vannier C, Hogrefe C, Marschner N, Grunwald V. First-line pazopanib in intermediate- and poor-risk patients with metastatic renal cell carcinoma: Final results of the FLIPPER trial. Int J Cancer. 2021 Feb 15;148(4):950-960. doi: 10.1002/ijc.33238. Epub 2020 Aug 18. PMID 32738823
- [Derived] Nel I, Gauler TC, Bublitz K, Lazaridis L, Goergens A, Giebel B, Schuler M, Hoffmann AC. Circulating Tumor Cell Composition in Renal Cell Carcinoma. PLoS One. 2016 Apr 21;11(4):e0153018. doi: 10.1371/journal.pone.0153018. eCollection 2016. PMID 27101285